CLINICAL TRIAL: NCT00371930
Title: Photodynamic Therapy for Permanent Hair Removal
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Jena (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1742-03/06
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Hypertrichosis; Hirsutism
MeSH Terms: conditions — Hypertrichosis; Hirsutism

INTERVENTIONS:
Procedure: application of a dye suspension followed by a laser intervention

SUMMARY:
24 test persons are treated with a dye suspension followed by a laser intervention. A decrease of hair density is expected.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60

Exclusion Criteria:

* anormal behavior
* pregnancy
* pathologic skin conditions
* medication that my interfere with the study
* allergy against the photosensitizer
* lack of compliance
* other reasons considered important by the investigator

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kaatz, Dr, Principal Investigator — FSU Jena
Locations (1):
- FSU Jena, Dept. of Dermatology, Jena, Thuringia, Germany